CLINICAL TRIAL: NCT00347815
Title: Pharmacokinetics and Pharmacodynamics of Buprenorphine After Intravenous Administration in Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of Buprenorphine in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish University of Pharmaceutical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROT-001-ML
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine the amount of buprenorphine and its metabolites in blood and urine after administration of 0.6 mg buprenorphine in healthy volunteers. Furthermore the purpose is to correlate the amount of buprenorphine in the blood with the effect on the ability to concentrate and coordinate.

ELIGIBILITY:
Inclusion Criteria:

healthy 18-40 years able to follow the protocol able to provide informed consent

Exclusion Criteria:

* Allergy to buprenorphine
* Mental illness
* Alcohol or drug abuse
* Chronic pain
* Daily use of analgesics
* Chronic medicinal treatment
* Treatment with corticosteroids
* Any use of medicine 48 hours before day of trial
* Smoker
* Blood donation within 3 months before day of trial
* Dementia
* Abnormal ECG
* Abnormal blood values:

Serum creatinine > 100 umol/l Serum haemoglobin < 8 mmol/L LDH < 105 U/L or > 255 U/L ASAT > 45 U/L ALAT > 70 U/L PP < 0.9 INR or > 1.1 INR Alkaline phosphatase < 35 U/L or > 275 U/L K+ < 3,5 mmol/L or > 5,0 mmol/L Na + < 136 mmol/L or > 146 mmol/

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-06; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Niels-Henrik Jensen, MD, Principal Investigator — Multidisciplinary Pain Centre, Herlev Hospital
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark